CLINICAL TRIAL: NCT05022056
Title: Impact of High-flow Nasal Oxygen During Awake Fiberoptic Bronchoscope Guided Intubation: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-0901
Record Dates: First submitted 2021-08-24; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Awake Fiberoptic Bronchoscope Guided Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective data collection. The aim of this study is to investigate impact of high-flow nasal oxygen on safety(lowest oxygen saturation), efficiency (intubation time, need for multiple attempts) in patients underwent awake fiberoptic bronchoscope guided intubation.

ELIGIBILITY:
Inclusion Criteria:

1.Patients who underwent awake fiberoptic bronchoscope guided intubation for surgery

Exclusion Criteria:

1. Cases in which other procedures (e.g. arterial line cannulation) were performed prior to endotracheal intubation after entering operation room
2. Patients with Incomplete records of oxygen saturation, attempt number, and time taken for awake intubation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent awake fiberoptic bronchoscope guided intubation for surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Intra-procedural lowest saturation | Intra-procedural lowest saturation
  Intra-procedural lowest saturation: lowest oxygen saturation on pulse oximetry during awake intubation
need for multiple attempts | Intra-procedural (need for multiple attempts : during awake intubation)
  need for multiple attempts : more than 2 attempts needed during awake intubation
time taken for awake intubation | Intra-procedural (Time taken for awake intubation: time from entering the operating room to completion of awake endotracheal intubation)
  Time taken for awake intubation: time from entering the operating room to completion of awake endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided